CLINICAL TRIAL: NCT05009433
Title: The Effect of Pre- and Postnatal High Intensity Interval Training and Moderate Intensity Continuous Training on Biological, Functional and Psychological Markers of Pregnancy Disorders and Non-communicable Diseases in Mothers and Offsprings
Brief Title: HIIT vs MICT During Pregnancy and Health and Birth Outcomes in Mothers and Children
Acronym: HIIT MAMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other); University of Gdansk (Other); Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1/KS/KF/DS2021
Record Dates: First submitted 2021-07-12; First posted 2021-08-17 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy; Postpartum; Childbirth; Health Status; Physical Fitness; Noncommunicable Diseases; Metabolism; Diabetes Mellitus, Gestational; Pregnancy Induced Hypertension; Body Composition; Back Pain; Pain Threshold; Biomechanics; Pelvic Floor Disorders; Urinary Incontinence; Cognitive Function; Depression; Anxiety
Keywords: Pregnant women; Prenatal care; Postpartum women; Postnatal care; Exercise; Physical activity; Exercise intervention; Educational intervention; Exercise test; High-intensity interval training; Moderate-intensity continuous training; Health Status; Physical fitness; Childbirth; Birth outcomes; Infant; Child
MeSH Terms: conditions — Noncommunicable Diseases; Diabetes, Gestational; Hypertension, Pregnancy-Induced; Back Pain; Pelvic Floor Disorders; Urinary Incontinence; Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study model is parallel in the two subgroups. The first subgroup consists of pregnant women who will be assigned to one of the three interventions: high intensity interval training program, moderate intensity continuous program or educational program on healthy lifestyle. The second subgroup will be age-matched nonpregnant women and they will be also assigned to the above three interventions. The pregnant women will be evaluated both in comparison to other pregnant women intervention groups and to the appropriate control non-pregnant groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the trial design and specificity of the interventions it is not possible to blind the study participants in terms of the allocation to the study groups. The HIIT and MICT groups will attend exercise sessions of high or moderate intesity, 3 times a week, while the comparative groups will not be subjected to any exercise intervention. However the data collectors and assessors will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pregnant HIIT group (Experimental): The high intensity interval training (HIIT) program will be implemented according to the World Health Organization guidelines on physical activity and sedentary behavior (2020) and on the recommendations on physical activity and exercise during pregnancy and postpartum period published by the American College of Obstetricians and Gynecologists (2020). The program will be also based on the "High-Intensity Interval Training for Cardiometabolic Disease Prevention" report by American College of Sports Medicine (2019). During the study, the participant will be under standard obstetric care on her own. She is obliged to inform her obstetric care provider about participation in the HIIT program and to provide feedback to the project coordinator as to possible recommendations of the obstetric care provider regarding the exercise.
  Interventions: Behavioral: High intensity interval training program for pregnant women
- Pregnant MICT group (Active Comparator): The moderate intensity continuous training (MICT) program will be implemented based on the World Health Organization guidelines on physical activity and sedentary behavior (2020) and on the recommendations on physical activity and exercise during pregnancy and postpartum period published by the American College of Obstetricians and Gynecologists (2020). During the study, the participant will be under standard obstetric care on her own. She is obliged to inform her obstetric care provider about participation in the MICT program and to provide feedback to the project coordinator as to possible recommendations of the obstetric care provider regarding the exercise.
  Interventions: Behavioral: Moderate intensity continuous training program for pregnant women
- Pregnant standard care group (Sham Comparator): During the study, the participant will be under standard obstetric care on her own. She is obliged to inform her obstetric care provider about participation in the HIIT Mama study and to provide feedback to the project coordinator as to possible contraindications to taking part in the study tests.
  Interventions: Behavioral: Standard obstetric care with extended education on healthy lifestyle
- Nonpregnant HIIT group (Experimental): The high intensity interval training (HIIT) program will be implemented according to the World Health Organization guidelines on physical activity and sedentary behavior (2020) and on the "High-Intensity Interval Training for Cardiometabolic Disease Prevention" report by American College of Sports Medicine (2019).
  During the study, the participant will be under standard health care on her own. She is obliged to inform her health care provider about participation in the HIIT Mama study and to provide feedback to the project coordinator as to possible contraindications to exercise or taking part in the study tests.
  Interventions: Behavioral: High intensity interval training program for nonpregnant women
- Nonpregnant MICT group (Active Comparator): The moderate intensity continuous training program will be implemented according to the World Health Organization guidelines on physical activity and sedentary behavior (2020).
  During the study, the participant will be under standard health care on her own. She is obliged to inform her health care provider about participation in the HIIT Mama study and to provide feedback to the project coordinator as to possible contraindications to exercise or taking part in the study tests.
  Interventions: Behavioral: Moderate intensity continuous training program for nonpregnant women
- Nonpregnant standard care group (Sham Comparator): During the study, the participant will be under standard health care on her own. She is obliged to inform her health care provider about participation in the HIIT Mama study and to provide feedback to the project coordinator as to possible contraindications to exercise or taking part in the study tests.
  Interventions: Behavioral: Standard health care with extended education on healthy lifestyle

INTERVENTIONS:
Behavioral: High intensity interval training program for pregnant women — Pregnant women will participate in 8-week HIIT cycles until the day of delivery, 3 times a week, in a volume of each session of 60 minutes. The main part (15-20 min) will be conducted in a form of high intensity intervals, approx. 85-90% of maximum exercise capacity. The intervals will consist of performing exercises for 30-60 seconds, alternating with a 30-60 second rest break, in the ratio of exercise time to rest 1:2, 1:1 or 2:1, according to the individual possibilities of the participant and taking into account the training progression and stage of pregnancy. The exercise intensity will be monitored with the use of heart rate monitors, the Borg Rating of Perceived Exertion (RPE) and the Talk Test.
  After birth, women will participate in 3-month HIIT cycles from the moment of achieving postpartum readiness to training until one year postpartum. Classes will be carried out stationary or online, depending on the pandemic situation and the availability of the woman.
  Other Names: HIIT during pregnancy
  Arms: Pregnant HIIT group
Behavioral: Moderate intensity continuous training program for pregnant women — Pregnant women will participate in 8-week MICT cycles until the day of delivery, 3 times a week, in a volume of each session of 60 minutes. The main part (20-25 min) will be conducted in a form of moderate intensity continuous exercise, of 70-80% of the maximum exercise capacity, e.g. in the form of high- and low-impact aerobics choreography with music. The sessions will also include resistance, neuromotor, body posture and flexibility exercises (25 min), breathing exercises, relaxation and visualization of pregnancy or childbirth (10 min). The exercise intensity will be monitored with the use of heart rate monitors, the Borg Rating of Perceived Exertion (RPE) and the Talk Test.
  After birth, women will participate in 3-month MICT cycles from the moment of achieving postpartum readiness to training until one year postpartum. Classes will be carried out stationary or online, depending on the pandemic situation and the availability of the woman.
  Other Names: MICT during pregnancy
  Arms: Pregnant MICT group
Behavioral: Standard obstetric care with extended education on healthy lifestyle — Pregnant women will get standard obstetric care according to the national law. They will attend educational sessions on a healthy lifestyle, physical activity in the perinatal period and selected aspects of pregnancy and motherhood. Educational classes will be conducted online in real time, at least once every two weeks, until one year postpartum.
  Arms: Pregnant standard care group
Behavioral: High intensity interval training program for nonpregnant women — Nonpregnant women will participate in 8-week HIIT cycles for a period of 8 months, 3 times a week, in a volume of each session of 60 minutes. The main part (15-20 min) will be conducted in a form of high intensity intervals, approx. 85-90% of maximum exercise capacity. The intervals will consist of performing exercises for 30-60 seconds, alternating with a 30-60 second rest break, in the ratio of exercise time to rest 1:2, 1:1 or 2:1, according to the individual possibilities of the participant and taking into account the training progression. The exercise intensity will be monitored with the use of heart rate monitors, the Borg Rating of Perceived Exertion (RPE) and the Talk Test.
  For the next 12 months of the project, women will participate in 3-month HIIT cycles. Classes will be carried out stationary or online, depending on the pandemic situation and the availability of the woman.
  Other Names: Lifetime HIIT
  Arms: Nonpregnant HIIT group
Behavioral: Moderate intensity continuous training program for nonpregnant women — Nonpregnant women will participate in 8-week MICT cycles for a period of 8 months, 3 times a week, in a volume of each session of 60 minutes. The main part (20-25 min) will be conducted in a form of moderate continuous intensity exercise, of 70-80% of the maximum exercise capacity, e.g. in the form of high- and low-impact aerobics choreography with music. The sessions will also include resistance, neuromotor, body posture and flexibility exercises (25 min), breathing exercises and relaxation (10 min). The exercise intensity will be monitored with the use of heart rate monitors, the Borg Rating of Perceived Exertion (RPE) and the Talk Test.
  For the next 12 months of the project, women will participate in 3-month MICT cycles. Classes will be carried out stationary or online, depending on the pandemic situation and the availability of the woman.
  Other Names: Lifetime MICT
  Arms: Nonpregnant MICT group
Behavioral: Standard health care with extended education on healthy lifestyle — Nonpregnant women will get standard health care according to the national law. They will attend educational sessions on a healthy lifestyle, physical activity and selected aspects of preparation to pregnancy and motherhood. Classes will be conducted online in real time, at least once every two weeks, for a period of 20 months.
  Arms: Nonpregnant standard care group

SUMMARY:
Regular exercise during pregnancy and postpartum leads to health benefits for mother and child. Inactivity during pregnancy and after delivery is now treated as risky behavior. Physically active pregnant women significantly less often suffer from, among others, gestational diabetes, excessive weight gain, lipids disorders, hypertension, preeclampsia, depressive symptoms, functional and structural disorders, including stress urinary incontinence, back pain or diastasis recti abdominis (DRA). Prenatal physical activity reduces the risk of premature delivery and miscarriage, fetal macrosomia, complications in labor or the risk of metabolic disorders in children.

High-intensity interval training (HIIT) has become one of the most popular trends in the fitness sector. The effectiveness of HIIT on a number of health indicators has been proven in various populations but limited data are available on HIIT during pregnancy.

The first hypothesis is that the HIIT, implemented during pregnancy and after childbirth, as a stronger exercise stimulus, will have a better impact on selected biological and psychological parameters of mothers, as well as on selected health parameters of their children, compared to the MICT (moderate intensity continuous training). Therefore, it promises better preventive effects on pregnancy complications and ailments as well as non-communicable diseases occurring in these populations. In the second hypothesis, it was assumed that HIIT and MICT implemented during pregnancy and after childbirth, tailored to the specific needs of the perinatal period, will not differ in the effectiveness of maintaining normal functional parameters in women, including prevention of urinary incontinence, back pain, DRA, etc.

Pregnant women who apply for the study will be divided into three groups: those attending the HIIT, MICT or educational programs. During the study, the participants will be under standard obstetric care. As comparative groups, non-pregnant women will be also recruited.

The investigators will collect data on selected biological, functional and psychological parameters in the study women at each trimester of pregnancy, during the puerperium and one year after childbirth. The data from the medical documentation on the course of childbirth and the assessment of the new-born, as well as the results of preventive examinations in the study women's children aged one, two, four and six years will be also analyzed.

ELIGIBILITY:
Inclusion Criteria:

Criteria: Inclusion Criteria:

For pregnant women:

1. course of pregnancy allowing participation in physical activities adapted to pregnant women
2. consent of the obstetric care provider to participate in the study tests and exercise classes;
3. taking part in all diagnostic and control tests to assess selected biological, functional and psychological parameters at each trimester of pregnancy, during the puerperium and one year after childbirth;
4. participant's consent to use data from the medical documentation on the course of childbirth and the assessment of the new-born, as well as the results of preventive examinations in children aged one, two, four and six, routinely performed according to the Polish pediatric care system;
5. availability to participate in classes three times a week until the day of delivery;
6. declaration of participation in postpartum classes at least once a week and self-completion of the exercise program according to written instructions prepared by the exercise specialist;
7. women can participate in the exercise programs regardless of their level of fitness or exercise capacity, as well as the level of motor skills (based on the diagnostic exercise tests, the exercise program will be tailored to the individual needs and capabilities of a woman).

For nonpregnant women:

1. nulliparous;
2. lack of diagnosed infertility and other disorders of the reproductive system;
3. taking part in all diagnostic and control tests to assess selected biological, functional and psychological parameters at indicated time points: before and after each of the 8-week exercise program during the first 8 months of the study and once every 3 months during the following twelve months of the study
4. declaration of availability to participate in exercise classes three times a week for the first 8 months of the program (attendance at least 80% is required);
5. declaration of participation in classes at least once a week and self-completion of the exercise program to the required 150 minutes of physical activity per week, according to the written guidelines prepared by the instructor, for the next 12 months of the program;
6. women can participate in the exercise program regardless of their level of fitness or exercise capacity, as well as the level of motor skills (based on the diagnostic exercise tests, the exercise program will be tailored to the individual needs and capabilities of a woman).

Exclusion Criteria for Pregnant and Nonpregnant Women:

1. contraindications to increased physical effort or to any of the diagnostic or control tests;
2. allergies to materials used during diagnostic and control tests (e.g. nickel present in steel plates of vaginal electrodes, disinfectants);
3. other conditions that, according to the researchers, will threaten the health or safety of the participants or will significantly affect the quality of the collected data.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in maternal oxygen consumption, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes from the baseline maternal oxygen consumption (VO2; ml/min), including the maximal oxygen consumption (VO2max) values in a progressive maximal exercise test on a cycloergometer with electronically regulated load, using stationary respiratory gas analyzer. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in maternal heart rate, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes from the baseline heart rate (HR; beats per minute), including the maximal HR values, in a progressive maximal exercise test on a cycloergometer with electronically regulated load, using heart rate monitor. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in systolic blood pressure, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes from the baseline maternal systolic blood pressure (SBP; mm Hg), in a progressive maximal exercise test on a cycloergometer with electronically regulated load, using electronic blood pressure monitor. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in diastolic blood pressure, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes from the baseline maternal diastolic blood pressure (DBP; mm Hg), in a progressive maximal exercise test on a cycloergometer with electronically regulated load, using electronic blood pressure monitor. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in blood glucose level, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in glucose levels (mg/dl) the blood samples will be taken on the day of the maximal exercise capacity test before the test (at fasting condition), immediately (approx. 1 min) after completion the test and approx. 40 min. after the test. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in triglycerides, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in triglycerides (TG; mg/dl) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in high-density lipoproteins, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in high-density lipoproteins (HDL; mg/dl) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in urea, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in urea levels (ml/dl), the study participants will collect urine samples to standard urine containers on the day of the maximal exercise capacity test before the test (at fasting condition), immediately after completion the test (up to 15 min) and approx. 60 min after the test. The investigators will analyze changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially related to renal function and changing with regular exercise in the perinatal period.
Changes in creatinine, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in creatinine levels (ml/dl), the study participants will collect urine samples to standard urine containers on the day of the maximal exercise capacity test before the test (at fasting condition), immediately after completion the test (up to 15 min) and approx. 60 min after the test. The investigators will analyze the changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially related to renal function and changing with regular exercise in the perinatal period.
Changes in maternal weight, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in maternal weight will be expressed in kilograms (kg). The investigators will analyze the changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in maternal Body Mass Index during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in Body Mass Index (BMI, kg/m2) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in maternal neuromuscular activity of pelvic floor muscles, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The neuromuscular activity of pelvic floor muscles (µV) will be evaluated with surface electromyography with a vaginal probe, in the condition of synergistic muscle relaxation. The investigators will analyze the changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to pelvic floor function and changing with regular exercise in the perinatal period.
Changes in the Incontinence Impact Questionnaire score, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The urinary incontinence symptoms will be assessed using the scale of incontinence impact on the quality of life based on the Incontinence Impact Questionnaire - short form (Uebersax et al., 1995; IIQ-7 score; minimum score: 0; maximum score: 100; higher scores mean worse outcome). The investigators will analyze the changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to pelvic floor function and changing with regular exercise in the perinatal period.
Changes in the Urogenital Distress Inventory score, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The pelvic floor disorders will be assessed using the scale based on the Urogenital Distress Inventory - short form questionnaire (Uebersax et al., 1995; UDI - 6 score; minimum score: 0; maximum score: 100; higher scores mean worse outcome). The investigators will analyze the changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to pelvic floor function and changing with regular exercise in the perinatal period.
Changes in the inter-rectus distance, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the inter-rectus distance (IRD, mm) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the center of pressure excursions (static balance), during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the excursions of the center of pressure (COP; mm) will be measured in standing position using a specialized force platform. The changes in the static balance will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in lumbar spine mobility, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the lumbar spine mobility (°) will be measured in standing position using specialized motion detectors and software. The changes lumbar spine mobility will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in cervical spine mobility, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the cervical spine mobility (°) will be measured in sitting position using specialized motion detectors and software. The changes lumbar spine mobility will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in foot loading, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in foot loading (kPa) will be measured in standing position using plantar pressure measurements platform and software. This outcome will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in spatiotemporal gait parameters: step length, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the step length (m) will be measured in walking using plantar pressure measurements platform and software. This outcome will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in spatiotemporal gait parameters: step width, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the step width (m) will be measured in walking using plantar pressure measurements platform and software. This outcome will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the hand grip strength, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The hand muscle strength (kg) will be assessed using the electronic hand grip dynamometer. The participant will perform the test separately for the right and left hands.
Changes in the pressure pain tolerance in the hand area, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The pressure pain tolerance (PTOL) will be assessed using a computerized pressure algometer in the hand area. The PTOL will be expressed in the value of applied pressure (kPa). The pain test will be performed before and immediately (up to 15 minutes) after the maximal exercise test on a cycloergometer.
  The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the pressure pain tolerance in the forearm area, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The pressure pain tolerance (PTOL) will be assessed using a computerized pressure algometer in the forearm area. The PTOL will be expressed in the value of applied pressure (kPa). The pain test will be performed before and immediately (up to 15 minutes) after the maximal exercise test on a cycloergometer. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in number of errors in the Stroop Interference test (version S8: congruent/incongruent), during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in reaction time based on the Stroop Interference test (version S8: congruent/incongruent), during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The time spent to complete each task, as well as the total time (s) to complete the Stroop Interference test will be assessed. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the Beck Depression Inventory - II score, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The occurrence and severity of depression symptoms using the scale of the Beck Depression Inventory - II (Beck et al., BDI -II score; minimum score: 0; maximum score: 63; higher scores mean worse outcome).The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the Fear of Childbirth questionnaire scores, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The fear of childbirth will be assessed using a scale based on the Fear of Childbirth scale questionnaire (Areskog et al., 1992; minimum score: 0; maximum score: 63; higher scores mean worse outcome). The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in cortisol level in hair, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The cortisol level (pg/mg) will be determined from a hair sample as a marker of permanent stress. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Complications of pregnancy: gestational diabetes mellitus | The data will be collected from the pregnant women groups before starting the intervention and after the completion of each training or educational cycle (each training or education cycle lasts 8 weeks) until childbirth.
  The incidence of gestational diabetes mellitus (GDM; % of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Complications of pregnancy: gestational hypertension | The data will be collected from the pregnant women groups before starting the intervention and after the completion of each training or educational cycle (each training or education cycle lasts 8 weeks) until childbirth.
  The incidence of gestational hypertension (GH; % of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Complications of pregnancy: preeclampsia | The data will be collected from the pregnant women groups before starting the intervention and after the completion of each training or educational cycle (each training or education cycle lasts 8 weeks) until childbirth.
  The incidence of preeclampsia (PE; % of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Complications of fetal development: fetal growth restriction | The data will be collected from the pregnant women groups before starting the intervention and after the completion of each training or educational cycle (each training or education cycle lasts 8 weeks) until childbirth.
  The incidence of fetal growth restriction (FGR; % of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Complications of fetal development: fetal macrosomia | The data will be collected from the pregnant women groups before starting the intervention and after the completion of each training or educational cycle (each training or education cycle lasts 8 weeks) until childbirth.
  The incidence of fetal macrosomia (FM; % of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: type of delivery | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The type of delivery (vaginal delivery, cesarean section, instrumental delivery; % of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: new-born's birth weight | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The new-born's birth weight (g) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: new-born's length | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The new-born's length (cm) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: APGAR score | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The APGAR score (the newborn's appearance, pulse, grimace, activity, and respiration score; minimum score: 0; maximum score: 10; higher scores mean better outcome) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childhood outcomes: changes in body weight | The data will be collected from the offsprings at one, two, four and six years of age.
  The changes in children's body weight (kg) will be analyzed in terms of pre- and postnatal physical activity patterns of their mothers and in relation to other selected parameters.
Childhood outcomes: changes in body height | The data will be collected from the offsprings at one, two, four and six years of age.
  The changes in children's body height (cm) will be analyzed in terms of pre- and postnatal physical activity patterns of their mothers and in relation to other selected parameters.
Childhood outcomes: changes in Body Mass Index | The data will be collected from the offsprings at one, two, four and six years of age.
  The changes in children's Body Mass Index (BMI; kg/m2) will be analyzed in terms of pre- and postnatal physical activity patterns of their mothers and in relation to other selected parameters.
Childhood outcomes: changes in systolic blood pressure | The data will be collected from the offsprings at one, two, four and six years of age.
  The changes in systolic blood pressure (SBP; mm Hg) in children will be analyzed in terms of pre- and postnatal physical activity patterns of their mothers and in relation to other selected parameters.
Childhood outcomes: changes in diastolic blood pressure | The data will be collected from the offsprings at one, two, four and six years of age.
  The changes in diastolic blood pressure (DBP; mm Hg) in children will be analyzed in terms of pre- and postnatal physical activity patterns of their mothers and in relation to other selected parameters.

SECONDARY OUTCOMES:
Changes in maternal carbon dioxide production, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes from the baseline carbon dioxide production (VCO2; ml/min) in a progressive maximal exercise test on a cycloergometer with electronically regulated load, using stationary respiratory gas analyzer. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in maternal minute ventilation, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes from the baseline maternal minute ventilation (VE; l/min), including the maximal minute ventilation (VEmax) values in a progressive maximal exercise test on a cycloergometer with electronically regulated load, using stationary respiratory gas analyzer. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in maternal respiratory rate, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes from the baseline maternal respiratory rate (RR; breaths per min) in a progressive maximal exercise test on a cycloergometer with electronically regulated load, using stationary respiratory gas analyzer. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in maternal exercise capacity, expressed in administered load, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in administered load (W) in a progressive maximal exercise test on a cycloergometer with electronically regulated load. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters.
Changes in total cholesterol, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in total cholesterol (TC; mg/dl) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in low-density lipoproteins, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in low-density lipoproteins (LDL; mg/dl) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in insulin concentration, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in insulin concentration (ng/ml), the samples will be taken on the day of the maximal exercise capacity test before the test (at fasting condition), immediately (approx. 1 min) after completion the test and approx. 40 min. after the test. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in irisin concentration, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in irisin concentration (ng/ml); the samples will be taken on the day of the maximal exercise capacity test before the test (at fasting condition), immediately (approx. 1 min) after completion the test and approx. 40 min. after the test. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in leptin concentration, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in leptin concentration (ng/ml); the samples will be taken on the day of the maximal exercise capacity test before the test (at fasting condition), immediately (approx. 1 min) after completion the test and approx. 40 min. after the test. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameter, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in adiponectin concentration, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in adiponectin concentration (ng/ml); the samples will be taken on the day of the maximal exercise capacity test before the test (at fasting condition), immediately (approx. 1 min) after completion the test and approx. 40 min. after the test. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameter, potentially related to metabolism and changing with regular exercise in the perinatal period.
Changes in albumin, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in albumin levels (mg/l), the study participants will collect urine samples to standard urine containers on the day of the maximal exercise capacity test before the test (at fasting condition), immediately after completion the test (up to 15 min) and approx. 60 min after the test. The serum albumin levels will be also determined. The investigators will analyze changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially related to renal function and changing with regular exercise in the perinatal period.
Changes in sodium, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in sodium levels (mmol/l), the study participants will collect urine samples to standard urine containers on the day of the maximal exercise capacity test before the test (at fasting condition), immediately after completion the test (up to 15 min) and approx. 60 min after the test. The serum sodium levels will be also determined. The investigators will analyze changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially related to renal function and changing with regular exercise in the perinatal period.
Changes in potassium, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  To assess the changes in potassium levels (mmol/l), the study participants will collect urine samples to standard urine containers on the day of the maximal exercise capacity test before the test (at fasting condition), immediately after completion the test (up to 15 min) and approx. 60 min after the test. The serum sodium levels will be also determined. The investigators will analyze changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially related to renal function and changing with regular exercise in the perinatal period.
Changes in maternal amount of body fat, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in maternal amount of body fat (%) will be assessed using the electrical bioimpedance method. The investigators will analyze changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in maternal lean body mass, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in maternal lean body mass (%) will be assessed using the electrical bioimpedance method. The investigators will analyze changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in maternal skeletal muscle mass, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in maternal skeletal muscle mass (%) will be assessed using the electrical bioimpedance method. The investigators will analyze changes in this parameters in terms of intervention mode and its relationship with other selected parameter, potentially changing with regular exercise in the perinatal period.
Changes in maternal body water, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  Changes in maternal skeletal body water (%) will be assessed using the electrical bioimpedance method. The investigators will analyze changes in this parameter in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the technique of voluntary pelvic floor muscle contraction, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The technique of voluntary pelvic floor muscle contraction (Szumilewicz et al. 2019; technique scores using 1-4 scale; minimum score: 1; maximum score: 4; higher scores mean better outcome) will be evaluated using surface electromyography with a vaginal probe. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to pelvic floor function and changing with regular exercise in the perinatal period.
Changes in maternal neuromuscular activity of pelvic floor muscles in contractions combining pelvic floor and synergistic muscles, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The neuromuscular activity of pelvic floor muscles (µV) will be evaluated with surface electromyography with a vaginal probe, in the condition of synergistic muscle activation.The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially related to pelvic floor function and changing with regular exercise in the perinatal period.
Changes in the Oswestry Disability Index, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will assess the occurrence and severity of back pain and its impact of the everyday life using the scale of the Oswestry Disability Index (Fairbank and Pynsent, 2000; ODI score; minimum score: 0; maximum score: 50; higher scores mean worse outcome). This outcome will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in spatiotemporal gait parameters: gait speed, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the gait speed (m/s) will be measured in walking using plantar pressure measurements platform and software. This outcome will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in spatiotemporal gait parameters: stride duration, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the stride duration (s) will be measured in walking using plantar pressure measurements platform and software. This outcome will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in spatiotemporal gait parameters: stance duration, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The changes in the stance duration (s) will be measured in walking using plantar pressure measurements platform and software. This outcome will be analyzed in terms of intervention mode and in relation to other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the SF-12 Physical Score, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will use the scale of Physical and Mental Health Status based on the Short Form-12 (SF-12) questionnaire (Gandek et al., 1998; PCS-12; minimum score: 24; maximum score: 57; higher scores mean better outcome). The Physical Score will be analyzed in relation to various intervention modes during the perinatal period.
Changes in the SF-12 Mental Score, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will use the scale of Physical and Mental Health Status based on the Short Form-12 (SF-12) questionnaire (Gandek et al., 1998; MCS-12; minimum score: 19; maximum score: 61; higher scores mean better outcome). The Mental Score will be analyzed in relation to various intervention modes during the perinatal period.
Changes in the Flourishing Scale score, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will use The Flourishing Scale (Diener et al., 2009; SF score; minimum score: 8; maximum score: 56; higher scores mean better outcome) to analyze the psychosocial aspects of participation in physical activity during the perinatal period.
Changes in the Fear of COVID-19 Scale score during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will use The Fear of COVID-19 Scale (Ahorsu et al., 2020; FCV-19S score; minimum score: 7; maximum score: 35; higher scores mean worse outcome)) will be assessed. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the pressure pain threshold in the hand area, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The pressure pain tolerance (PPT) will be assessed using a computerized pressure algometer in the hand area. The PPT will be expressed in the value of applied pressure (kPa). The pain test will be performed before and immediately (up to 15 minutes) after the maximal exercise test on a cycloergometer. The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in the pressure pain threshold in the forearm area, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The pressure pain tolerance (PPT) will be assessed using a computerized pressure algometer in the forearm area. The PPT will be expressed in the value of applied pressure (kPa). The pain test will be performed before and immediately (up to 15 minutes) after the maximal exercise test on a cycloergometer.
  The investigators will analyze changes in this outcome in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Changes in serum cortisol level, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will analyze the changes in serum cortisol level (ng/ml) induced by the maximal exercise test and the intervention mode, and its relationship with other selected parameters, potentially related to depression, anxiety and stress levels and changing with regular exercise in the perinatal period.
Changes in serum oxytocin level, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will analyze the changes in serum oxytocin level (ng/ml) induced by the maximal exercise test and the intervention mode, and its relationship with other selected parameters, potentially related to depression, anxiety and stress levels and changing with regular exercise in the perinatal period.
Changes in serum dopamine level, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will analyze the changes in serum dopamine level (ng/ml) induced by the maximal exercise test and the intervention mode, and its relationship with other selected parameters, potentially related to depression, anxiety and stress levels and changing with regular exercise in the perinatal period.
Changes in serum adrenaline level, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will analyze the changes in serum adrenaline level (ng/ml) induced by the maximal exercise test and the intervention mode, and its relationship with other selected parameters, potentially related to depression, anxiety and stress levels and changing with regular exercise in the perinatal period.
Changes in serum serotonin level, during and after pregnancy | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will analyze the changes in serum serotonin level (ng/ml) induced by the maximal exercise test and the intervention mode, and its relationship with other selected parameters, potentially related to depression, anxiety and stress levels and changing with regular exercise in the perinatal period.
Childbirth parameters: gestational age at birth | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The gestational age at birth (weeks) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: length of labor | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The length of labor (hours and minutes) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: induction of labor | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The rate of induction of labor (% of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: episiotomy | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The rate of episiotomy (% of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: perineal lacerations | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The incidence of perineal lacerations (% of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: the use of anesthetics | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The rate of anesthetics use (% of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: labor complications | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The incidence of labor complications (% of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childbirth parameters: neonatal intensive care unit | The data will be collected from the pregnant women groups in the first two months after their childbirth.
  The incidence of neonatal intensive care unit (NICU; % of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.
Childhood outcomes: changes in percentage of body fat | The data will be collected from the offsprings at one, two, four and six years of age.
  The changes in amount of body fat in children (%) will be analyzed in terms of pre- and postnatal physical activity patterns of their mothers and in relation to other selected parameters.
Covid-19 disease | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The incidence of Covid-19 disease (% of the study group) will be analyzed in terms of intervention mode and its relationship with other selected parameters, potentially changing with regular exercise in the perinatal period.

OTHER OUTCOMES:
The level of physical activity based on the International Physical Activity Questionnaire | Before starting the intervention and after the completion of each training or educational cycle (during the first 8 months or until birth each training or education cycle lasts 8 weeks; during the next 12 months each cycle lasts 3 months).
  The investigators will use the International Physical Activity Questionnaire to calculate IPAQ score (minimum score: 0; maximum score: not specified; higher scores mean better outcome) to determine the participants' levels of physical activity prior to enrollment in the study and during the study.
Ten Item Personality Inventory score | Before starting the intervention.
  The investigators will use the Ten Item Personality Inventory (Gosling et al., 2003; TIPI scores; minimum score: 2; maximum score: 14; the higher the score, the greater the intensity of the personality traits) to analyze the psychosocial determinants of participation in physical activity during the perinatal period.
Life Orientation Test - Revised score | Before starting the intervention.
  The investigators will use the optimism versus pessimism scale based on the Life Orientation Test - Revised (Scheier et al., 1994; LOT-R score; minimum score: 6; maximum score: 24; the higher the score, the higher level of optimism) to analyze the psychosocial determinants of participation in physical activity during the perinatal period.
The Fat mass and obesity-associated (FTO) gene polymorphism | Before starting the intervention.
  The Fat mass and obesity-associated (FTO) gene polymorphism will be analyzed as a determinant of the incidence of metabolic disorders during pregnancy and postpartum, in relation to different patterns of physical activity and other selected parameters.
The Mu-Opioid Receptor Genetic Polymorphism (OPRM1) | Before starting the intervention.
  The Mu-Opioid Receptor Genetic Polymorphism (OPRM1) will be analyzed as a determinant of pain perception during pregnancy, labor and postpartum, in relation to different patterns of physical activity and other selected parameters.
The serotonin transporter (5-HTTLPR) polymorphism | Before starting the intervention.
  The serotonin transporter (5-HTTLPR) polymorphism will be analyzed as a determinant of depressive symptoms and anxiety during pregnancy and postpartum, in relation to different patterns of physical activity and other selected parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Anna N Szumilewicz, Assoc. Prof., Principal Investigator — Gdansk University of Physical Activity and Sport
Locations (1):
- Laboratory of Physical Effort and Genetics in Sport at Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results reported in publications will be available to other researchers. All procedures will be conducted in accordance with the Regulation (2016/679) of the European Parliament and of the Council of 27 April 2016 on the protection of individuals with regard to the processing of personal data and on the free movement of such data and repealing Directive 95/46 / EC. Each data set will be linked to a given research task description, the methods used to generate the data, the period of time data were collected and whether the data have been updated. The data will be stored in the standard file formats, such as MS Excel (.xlsx), MS Word (.docx), Comma Separated Values (.csv), Portable Document Format (.pdf), Joint Photographic Experts Group (.jpg), Tagged Image File Format (.tiff). Transformation of the high-resolution images may be necessary prior to data sharing. No further manipulation of these files is necessary.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available 6 months after publication, for a period of 10 years.
Access Criteria: All data published in peer-reviewed scientific journals will be made available to all interested researchers and preserved long-term. Data will be made available via open-access repository following the acceptance of the scientific journal, publishing the study reports. The process for gaining access to non-publicly accessible data will be straightforward and involve email communication to the Principal Investigator. We expect no embargo periods for political/commercial/patent or publishing process reasons. The URL for the data repository will be shared as soon as it is ready.

REFERENCES:
- [Background] Bo K, Artal R, Barakat R, Brown W, Davies GA, Dooley M, Evenson KR, Haakstad LA, Henriksson-Larsen K, Kayser B, Kinnunen TI, Mottola MF, Nygaard I, van Poppel M, Stuge B, Khan KM. Exercise and pregnancy in recreational and elite athletes: 2016 evidence summary from the IOC expert group meeting, Lausanne. Part 1-exercise in women planning pregnancy and those who are pregnant. Br J Sports Med. 2016 May;50(10):571-89. doi: 10.1136/bjsports-2016-096218. No abstract available. PMID 27127296
- [Background] Bo K, Artal R, Barakat R, Brown W, Dooley M, Evenson KR, Haakstad LAH, Larsen K, Kayser B, Kinnunen TI, Mottola MF, Nygaard I, van Poppel M, Stuge B, Davies GAL; IOC Medical Commission. Exercise and pregnancy in recreational and elite athletes: 2016 evidence summary from the IOC expert group meeting, Lausanne. Part 2-the effect of exercise on the fetus, labour and birth. Br J Sports Med. 2016 Nov;50(21):1297-1305. doi: 10.1136/bjsports-2016-096810. Epub 2016 Oct 12. PMID 27733352
- [Background] Bo K, Artal R, Barakat R, Brown WJ, Davies GAL, Dooley M, Evenson KR, Haakstad LAH, Kayser B, Kinnunen TI, Larsen K, Mottola MF, Nygaard I, van Poppel M, Stuge B, Khan KM; IOC Medical Commission. Exercise and pregnancy in recreational and elite athletes: 2016/17 evidence summary from the IOC Expert Group Meeting, Lausanne. Part 3-exercise in the postpartum period. Br J Sports Med. 2017 Nov;51(21):1516-1525. doi: 10.1136/bjsports-2017-097964. Epub 2017 Jun 22. No abstract available. PMID 28642221
- [Background] Davenport MH, Ruchat SM, Poitras VJ, Jaramillo Garcia A, Gray CE, Barrowman N, Skow RJ, Meah VL, Riske L, Sobierajski F, James M, Kathol AJ, Nuspl M, Marchand AA, Nagpal TS, Slater LG, Weeks A, Adamo KB, Davies GA, Barakat R, Mottola MF. Prenatal exercise for the prevention of gestational diabetes mellitus and hypertensive disorders of pregnancy: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1367-1375. doi: 10.1136/bjsports-2018-099355. PMID 30337463
- [Background] Davenport MH, Nagpal TS, Mottola MF, Skow RJ, Riske L, Poitras VJ, Jaramillo Garcia A, Gray CE, Barrowman N, Meah VL, Sobierajski F, James M, Nuspl M, Weeks A, Marchand AA, Slater LG, Adamo KB, Davies GA, Barakat R, Ruchat SM. Prenatal exercise (including but not limited to pelvic floor muscle training) and urinary incontinence during and following pregnancy: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1397-1404. doi: 10.1136/bjsports-2018-099780. PMID 30337466
- [Background] Davenport MH, Ruchat SM, Sobierajski F, Poitras VJ, Gray CE, Yoo C, Skow RJ, Jaramillo Garcia A, Barrowman N, Meah VL, Nagpal TS, Riske L, James M, Nuspl M, Weeks A, Marchand AA, Slater LG, Adamo KB, Davies GA, Barakat R, Mottola MF. Impact of prenatal exercise on maternal harms, labour and delivery outcomes: a systematic review and meta-analysis. Br J Sports Med. 2019 Jan;53(2):99-107. doi: 10.1136/bjsports-2018-099821. Epub 2018 Oct 18. PMID 30337349
- [Background] Davenport MH, McCurdy AP, Mottola MF, Skow RJ, Meah VL, Poitras VJ, Jaramillo Garcia A, Gray CE, Barrowman N, Riske L, Sobierajski F, James M, Nagpal T, Marchand AA, Nuspl M, Slater LG, Barakat R, Adamo KB, Davies GA, Ruchat SM. Impact of prenatal exercise on both prenatal and postnatal anxiety and depressive symptoms: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1376-1385. doi: 10.1136/bjsports-2018-099697. PMID 30337464
- [Background] Perales M, Valenzuela PL, Barakat R, Cordero Y, Pelaez M, Lopez C, Ruilope LM, Santos-Lozano A, Lucia A. Gestational Exercise and Maternal and Child Health: Effects until Delivery and at Post-Natal Follow-up. J Clin Med. 2020 Jan 31;9(2):379. doi: 10.3390/jcm9020379. PMID 32023833
- [Background] Physical Activity and Exercise During Pregnancy and the Postpartum Period: ACOG Committee Opinion, Number 804. Obstet Gynecol. 2020 Apr;135(4):e178-e188. doi: 10.1097/AOG.0000000000003772. PMID 32217980
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Batrakoulis A. European survey of fitness trends for 2020. ACSM's Health & Fitness Journal. 2019;23(6):28-35. PubMed PMID: 141012112.
- [Background] Campbell WW, Kraus WE, Powell KE, Haskell WL, Janz KF, Jakicic JM, Troiano RP, Sprow K, Torres A, Piercy KL, Bartlett DB; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. High-Intensity Interval Training for Cardiometabolic Disease Prevention. Med Sci Sports Exerc. 2019 Jun;51(6):1220-1226. doi: 10.1249/MSS.0000000000001934. PMID 31095079
- [Background] Yeh SW, Lin LF, Chen HC, Huang LK, Hu CJ, Tam KW, Kuan YC, Hong CH. High-intensity functional exercise in older adults with dementia: A systematic review and meta-analysis. Clin Rehabil. 2021 Feb;35(2):169-181. doi: 10.1177/0269215520961637. Epub 2020 Oct 11. PMID 33040592
- [Background] Lavin-Perez AM, Collado-Mateo D, Mayo X, Humphreys L, Liguori G, James Copeland R, Del Villar Alvarez F, Jimenez A. High-intensity exercise to improve cardiorespiratory fitness in cancer patients and survivors: A systematic review and meta-analysis. Scand J Med Sci Sports. 2021 Feb;31(2):265-294. doi: 10.1111/sms.13861. Epub 2020 Nov 5. PMID 33098219
- [Background] Songstad NT, Kaspersen KH, Hafstad AD, Basnet P, Ytrehus K, Acharya G. Effects of High Intensity Interval Training on Pregnant Rats, and the Placenta, Heart and Liver of Their Fetuses. PLoS One. 2015 Nov 13;10(11):e0143095. doi: 10.1371/journal.pone.0143095. eCollection 2015. PMID 26566220
- [Background] Ong MJ, Wallman KE, Fournier PA, Newnham JP, Guelfi KJ. Enhancing energy expenditure and enjoyment of exercise during pregnancy through the addition of brief higher intensity intervals to traditional continuous moderate intensity cycling. BMC Pregnancy Childbirth. 2016 Jul 15;16(1):161. doi: 10.1186/s12884-016-0947-3. PMID 27417194
- [Background] Szumilewicz A, Worska A, Santos-Rocha R, Oviedo-Caro M. Evidence-based and practice-oriented guidelines for exercising during pregnancy. In: Santos-Rocha R, editor. Exercise and sporting activity during pregnancy Evidence-based guidelines. Cham: Springer International Publishing; 2019. p. 157-81.
- [Background] Santos-Rocha R, Gutiérrez I, Szumilewicz A, Pajaujiene S. Exercise testing and prescription for pregnant women. In: Santos-Rocha R, editor. Exercise and sporting activity during pregnancy: evidence-based guidelines. Cham: Springer International Publishing; 2019. p. 183-230.
- [Background] Szumilewicz A, Santos-Rocha R. Exercise selection and adaptation during pregnancy. In: Santos-Rocha R, editor. Exercise and sporting activity during pregnancy Evidence-based guidelines. Cham: Springer International Publishing; 2019. p. 231-308.
- [Background] Szumilewicz A, Worska A, Piernicka M, Kuchta A, Kortas J, Jastrzebski Z, Radziminski L, Jaworska J, Micielska K, Ziemann E. The Exercise-Induced Irisin Is Associated with Improved Levels of Glucose Homeostasis Markers in Pregnant Women Participating in 8-Week Prenatal Group Fitness Program: A Pilot Study. Biomed Res Int. 2017;2017:9414525. doi: 10.1155/2017/9414525. Epub 2017 Oct 31. PMID 29226153
- [Background] Szumilewicz A, Worska A, Piernicka M, Kuchta A, Jastrzebski Z, Radziminski L, Kozlowska M, Micielska K, Ziemann E. Acute Postexercise Change in Circulating Irisin Is Related to More Favorable Lipid Profile in Pregnant Women Attending a Structured Exercise Program and to Less Favorable Lipid Profile in Controls: An Experimental Study with Two Groups. Int J Endocrinol. 2019 Feb 28;2019:1932503. doi: 10.1155/2019/1932503. eCollection 2019. PMID 30944566
- [Background] Szumilewicz A, Dornowski M, Piernicka M, Worska A, Kuchta A, Kortas J, Bludnicka M, Radziminski L, Jastrzebski Z. High-Low Impact Exercise Program Including Pelvic Floor Muscle Exercises Improves Pelvic Floor Muscle Function in Healthy Pregnant Women - A Randomized Control Trial. Front Physiol. 2019 Jan 30;9:1867. doi: 10.3389/fphys.2018.01867. eCollection 2018. PMID 30761019
- [Background] Szumilewicz A, Kuchta A, Kranich M, Dornowski M, Jastrzebski Z. Prenatal high-low impact exercise program supported by pelvic floor muscle education and training decreases the life impact of postnatal urinary incontinence: A quasiexperimental trial. Medicine (Baltimore). 2020 Feb;99(6):e18874. doi: 10.1097/MD.0000000000018874. PMID 32028397
- [Background] Budnik-Przybylska D, Laskowski R, Pawlicka P, Anikiej-Wiczenbach P, Lada-Masko A, Szumilewicz A, Makurat F, Przybylski J, Soya H, Kazmierczak M. Do Physical Activity and Personality Matter for Hair Cortisol Concentration and Self-Reported Stress in Pregnancy? A Pilot Cross-Sectional Study. Int J Environ Res Public Health. 2020 Nov 1;17(21):8050. doi: 10.3390/ijerph17218050. PMID 33139602
- [Background] Santos-Rocha R, Szumilewicz A, Perales M, Pajaujiene S. EuropeActive Standards EQF Level 5 - Pregnancy and Postnatal Exercise Specialist. Brussels: EuropeActive; 2016.
- [Derived] Sun J, Radziminski L, Santos-Rocha R, Szumilewicz A. High-intensity interval training is an effective exercise mode to maintain normal blood pressure during pregnancy: a randomized control trial. Sci Rep. 2024 Nov 14;14(1):27975. doi: 10.1038/s41598-024-79552-3. PMID 39543304
- [Derived] Wilczynska D, Walczak-Kozlowska T, Radziminski L, Oviedo-Caro MA, Santos-Rocha R, Szumilewicz A. Can we hit prenatal depression and anxiety through HIIT? The effectiveness of online high intensity interval training in pregnant women during the COVID-19 pandemic: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Dec 22;14(1):215. doi: 10.1186/s13102-022-00610-2. PMID 36550564